CLINICAL TRIAL: NCT06528600
Title: A Randomized, Double-Blind, Active Controlled, Multi-Center, Non- Inferiority Study of One-injection of Hymovis ONE (32 mg/4ml) Against Currently Approved 1-injection Regimen of Monovisc in Symptomatic Relief of Osteoarthritis of the Knee
Brief Title: Comparative Study of Two Hyaluronic Acid Formulation in the Management of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EQE9-18-01
Record Dates: First submitted 2024-05-08; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized (1:1 allocation Hymovis ONE®: Monovisc™), double-blind, active comparator-controlled, non-inferiority study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hymovis One (Experimental): Treatment with 4 mL of Hymovis ONE® in the Intra-articular space
  Interventions: Device: Hymovis ONE
- Monovisc (Active Comparator): Treatment with 4 mL of Monovisc™ in the Intra-articular space
  Interventions: Device: Monovisc

INTERVENTIONS:
Device: Hymovis ONE — Single injection of Hymovis ONE®, a sodium hyaluronate formulation, for the treatment of pain from osteoarthritis (OA) of the knee in patients who have not responded to non-pharmacological therapies or analgesic regimens
  Arms: Hymovis One
Device: Monovisc — Single injection of Monovisc™ a sodium hyaluronate formulation, for the treatment of pain from osteoarthritis (OA) of the knee in patients who have not responded to non-pharmacological therapies or analgesic regimens
  Arms: Monovisc

SUMMARY:
The objective of this randomized, double-blind, active-controlled, non-inferiority study is to compare the effectiveness and safety of a single injection of Hymovis ONE®, a sodium hyaluronate formulation, to Monovisc™, another sodium hyaluronate formulation, for the treatment of pain from osteoarthritis (OA) of the knee in patients who have not responded to non-pharmacological therapies or analgesic regimens. This study consists of a 2-week period for screening, one baseline treatment visit, and a 26- week evaluation phase. Subjects will be randomized to receive a single intra-articular (IA) injection of either Hymovis ONE® or Monovisc™ into the knee using an 18-20 gauge needle.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, active comparator-controlled, non-inferiority study to assess the efficacy and safety of a single injection of Hymovis ONE® for the relief of pain in subjects with OA of the knee by establishing its non-inferiority to Monovisc™.

The entire study will last approximately 19 months. Patients will participate in the study for approximately 28 weeks (from screening to the last visit).

The study is designed to compare the effectiveness and safety of a single injection of Hymovis ONE® to a single injection of Monovisc™. Both products are high molecular weight HA preparations, specifically sodium hyaluronate from bacterial fermentation, supplied sterile as a single dose of 4 ml in a 5 ml syringe.

Subjects will undergo an evaluation consisting of a thorough discussion of medical history, demographics, followed by a physical examination and vital signs (blood pressure and heart rate) measurement.

The evaluation of their activity level through the Tegner activity level scale, a graduated list of ADLs, recreation, and competitive sports will be performed. The patient is asked to select the level of participation that best describes their current level of activity through an Investigator's interview. The Tegner activity level scale is filled in by Investigator.

In this study, one single IA injection of Hymovis ONE® or Monovisc™ will be performed at the investigational site, under the tight supervision of an experienced treating specialist. Therefore, there are no expected risks of misuse in the administration of the investigational products according to treatment schedule defined in the study protocol. Furthermore, the use of only one IA injection should further contribute to limit the risk of adverse effects. Therefore, it is expected that benefits from participation in this study will outweigh the potential risks.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male subjects ≥ 40 and ≤ 75 years of age
2. Body mass index (BMI) ≥20 and <35 kg/m2
3. Tegner score ≥3
4. Subjects with primary knee OA of the medial or lateral femorotibial compartment with symptoms at screening and for at least 3 months prior to screening according to American College of Rheumatology (ACR) criteria and who have not responded to conservative non-pharmacologic treatment or simple analgesic regimens
5. Subjects with Kellgren-Lawrence (K-L) radiological grade 2 or 3 in the target knee
6. Subjects with at least one X-Ray image of the target knee taken at screening or within 6 months prior to the screening.
7. Subjects with OA pain intensity meeting the criteria below:

   * Subjects demonstrating at both the screening (V0) and the baseline (V1) visit, pain intensity in the target knee of 2 - 3 and in the contralateral knee 0 as measured by the WOMAC LK3.1 A1 Pain subscale (walking on a flat surface)
8. Willingness to discontinue oral and topical analgesics including NSAIDs and accept "rescue" paracetamol as the only medicine for joint pain prior to the injection and throughout the study. "Rescue" medication will be discontinued 24 hours before any study visit
9. Subjects able to understand and willing and able to comply with study procedures
10. Subjects able to provide informed consent
11. If female of childbearing potential, must have a negative pregnancy test at screening and agree to use a reliable form of contraception throughout the study*.

Note: To be considered of non-childbearing potential, females must be surgically sterile or postmenopausal for at least 1 year.

*Highly effective birth control methods include: combined hormonal contraception containing estrogen and progestogen) associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD); intrauterine ormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence.

Exclusion Criteria:

1. Inability to perform a 50-foot walk test
2. Subjects with secondary (post-traumatic) knee OA of the target joint
3. Subjects with K-L radiological grade 1 or 4 in the target knee
4. Subjects with known X-ray findings of acute fractures, severe loss of bone density, avascular necrosis, and /or severe bone or joint deformity in the target knee
5. Clinically apparent tense effusion of the target knee on examination (determined by either a positive bulge sign or ballottement of the patella (patellar tap))
6. Subjects with osteonecrosis of either knee
7. Subjects with a history of knee joint replacement or arthroplasty of the target knee
8. Subjects with a history of arthroscopy of the target knee in the past 6 months
9. Subjects with a history of osteotomy or surgery of the target or contralateral knee and any other weight-bearing joint that would have interfered with knee assessment
10. Subjects with acute, recurrent synovitis, or any inflammatory conditions in the target knee
11. Subjects with any significant injury to the target knee in the last 6 months (as per Investigator judgment)
12. Subjects with any musculoskeletal condition affecting the target knee that would impair the proper assessment of the

    Investigational Medical Device (IMD) performance in the target knee as assessed by the Investigator such as:
    1. severe varus/valgus deformity (>15°)
    2. predominantly patellofemoral pain syndrome
13. Subjects with health condition associated with pain which may interfere with study variables evaluation
14. Subjects with a known history or present evidence of conditions which may affect the target knee assessments, like rheumatic disease, lupus arthropathy, infective or metabolic joint diseases; recurrent clinical chondrocalcinosis; crystal arthropathies; osteoarticular pathologies differing from arthrosis; acromegaly; haemochromatosis; Wilson's disease; primary osteochondromatosis; heritable disorders; collagen gene mutations
15. Subjects with gout or calcium pyrophosphate (pseudogout) diseases of the target knee with flare-ups within 6 months prior to screening
16. Subjects with fibromyalgia, pes anserine bursitis, lumbar radiculopathy and/or neurogenic or vascular claudication
17. Subject with significant anterior knee pain due to the diagnosed isolated patellar-femoral syndrome or chondromalacia in the target knee
18. Subjects with symptomatic OA of the hips, spine or ankle that interferes with the evaluation of the target knee
19. Subjects with venous or lymphatic stasis in the relevant limb
20. Subjects with a history of the following treatments:

    1. IA corticosteroids in any joints in the past 3 months
    2. Systemic (both oral and parenteral) and topical corticosteroids at the target knee in the past 30 and 90 days, respectively
    3. Topical anti-inflammatory agents and analgesics applied at the target knee in the past 48 hours
    4. Viscosupplementation with hyaluronic acid or joint-lavage in the target knee in the past 6 months
    5. Physical therapy started in the past 3 months in the target knee. Subjects having started a physical therapy from more than 3 months can take part in the study
    6. Change in the dosage of symptomatic slow-acting supplements for OA such as glucosamine, chondroitin sulfate, diacerhein, or other supplements such as avocado or soya extracts, etc. in the last month
    7. Chronic or recurrent use of narcotic analgesics
21. Subjects with a history of chronic or recurrent use of NSAIDs/analgesics/narcotics because of diseases different from OA of the target knee
22. Subjects treated with agents which alter the perception of pain such as hypnotics, muscle relaxants, anxiolytics if the intake has started less than 8 days before screening
23. Subjects with a history of recurrent severe allergic or immune-mediated reactions or other immune disorders
24. Subjects with vascular insufficiency of lower limbs or peripheral neuropathy severe enough to interfere
25. Subjects with active liver disease
26. Subjects with any clinically significant laboratory values which, based on investigator judgment and subject clinical history, may affect study evaluation
27. Subjects who currently use heparin or anti-vitamin K (e. g. crystalline warfarin) anticoagulant therapy
28. Subjects with infections, wounds, bruising, disease or trauma in the area of the injection site or joint
29. Subjects with suspected or known history of hypersensitivity to paracetamol, lidocaine, hyaluronic acid or to hyaluronate preparations or gram-positive bacterial proteins
30. Subjects with any surgical procedures scheduled in the next 6 months
31. Subjects who have participated in a clinical study or investigation in the last 3 months
32. Pregnant or lactating women, and women of childbearing potential unwilling to use adequate contraception and conduct a pregnancy test at screening.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Pain relief compared to baseline | week 12
  Change From Baseline (CFB) in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) LK3.1 A1 Pain subscale (walking on a flat surface) score

SECONDARY OUTCOMES:
Patient respons to treatment | Week 12 and 26
  "Patient Success" is defined by OMERACT-OARSI criteria:
  (1) improvement in pain or physical function ≥50% and an absolute change ≥20; or (2) improvement of ≥20% with an absolute change of≥ 10 in at least two of the following three categories: pain, physical function, and patient's global assessment
Pain relief compared to baseline | Week 26
  Change from Baseline (CFB) in the Pain subscale in WOMAC LK3.1
Joint Stiffness compared to baseline | Week 26
  Change from Baseline (CFB) in the WOMAC LK3.1 Stiffness
Joint Function compared to baseline | Week 26
  Change from Baseline (CFB) in the WOMAC LK3.1 Function
Patient quality of life | Weeks 4,12 and 26
  Evaluation through SF-12 questionnaire
Patient Global Assessment (PGA) | Weeks 4,12 and 26
  Evaluation of disease severity measured by patient using a 0-100 Visual Analogue Scale (VAS) as a Change From Baseline
Clinical Observer Global Assessment (COGA) | Weeks 4,12 and 26
  Evaluation of disease severity measured by clinician using a 0-100 Visual Analogue Scale (VAS) as a Change From Baseline
Rescue paracetamol use | up to 26 weeks
  evaluation of paracetamol consumption during the study duration through a patient diary
Safety of the treatment. Number of patient with treatment related adverse events | up to 26 weeks
  Safety evaluation by tracking the number of adverse events correlated to treatment at each visit

CONTACTS AND LOCATIONS:
Locations (19):
- Italy (19):
  - Fondazione Poliambulanza , Istituto Ospedaliero UO di Ortopedia e Traumatologia, Brescia, BS
  - ASST Valcamonica U.O.C. Ortopedia, Esine, BS
  - A.O.R.N. S. Anna e S. Sebastiano U.O.C. Ortopedia e Traumatologia, Caserta, CE
  - U.O. Ortopedia e Traumatologia Casa di Cura, Maddaloni, CE
  - A.O. Ospedale Santa Croce e Carle S.C. Ortopedia e Traumatologia, Cuneo, CN
  - Ospedale S. Maria Borgo Val di Taro - AUSL Parma U.O. Ortopedia e Traumatologia, Borgo Val di Taro, PR
  - Azienda Ospedaliero-Universitaria di Parma U.O. Clinica Ortopedica, Parma, PR
  - Fondazione IRCCS Policlinico San Matteo Pavia U.O.C. Ortopedia e Traumatologia, Pavia, PV
  - Policlinico universitario Campus Biomedico, Roma, RO
  - Ospedale San Giovanni Calibita Fatebenefratelli - Isola Tiberina U.O.C. di Ortopedia e Traumatologia, Roma, RO
  - Ospedale Santo Spirito in Sassia - ASL Roma 1 Ortopedia e Traumatologia, Roma, RO
  - A.O. Città della Salute e della Scienza - Presidio CTO (Centro Traumatologico Ortopedico) S.C. Ortopedia e Traumatologia 1 U, Torino, TO
  - AOU Città della Salute e della Scienza di Torino -Ospedale Molinette S.C. Medicina Fisica e Riabilitazione U Dip. Ortopedia Traumatologia e Riabilitazione, Torino, TO
  - Presidio Sanitario Ospedale Cottolengo Ortopedia, Torino, TO
  - Azienda ULSS 2 Marca Trevigiana - Ospedale di Conegliano U.O.C. Ortopedia e Traumatologia, Conegliano, TV
  - A.O. Ospedale Cardarelli I Ortopedia, Napoli
  - AOU Federico II Napoli UOC Ortopedia e Traumatologia, Napoli
  - P.O. Ospedale del Mare ASL 1 Napoli U.O.C. Ortopedia, Napoli
  - A.O.U. " Maggiore della Carità" S.C. di Ortopedia e Traumatologia, Novara

IPD SHARING:
Plan to Share IPD: No